CLINICAL TRIAL: NCT02097069
Title: Different Effects of Inositol Stereoisomers on Insulin Sensitivity in Women With Gestational Diabetes
Brief Title: Inositol Stereoisomers to Treat Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Ester Vitacolonna, Professor Ester Vitacolonna, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITA01
Record Dates: First submitted 2014-02-27; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus; Myo-inositol; D-chiro-inositol; Insulin resistance
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Folic Acid; Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Subgroup A (Other): folic acid 400 mcg/day
  Interventions: Dietary Supplement: Folic acid
- Subgroup B (Experimental): myo-inositol 2000 mg twice a day
  Interventions: Dietary Supplement: Myo-inositol
- Subgroup C (Experimental): D-chiro-inositol 250 mg twice a day
  Interventions: Dietary Supplement: D-Chiro-inositol
- Subgroup D (Experimental): Myo-inositol plus D-chiro inositol 550mg/13,8 mg twice a day
  Interventions: Dietary Supplement: Myo-inositol plus D-chiro inositol

INTERVENTIONS:
Dietary Supplement: Folic acid — Folic acid 400 mcg/day
  Arms: Subgroup A
Dietary Supplement: Myo-inositol — myo-inositol 2000 mg twice a day
  Arms: Subgroup B
Dietary Supplement: D-Chiro-inositol — D-chiro inositol 250 mg twice a day
  Arms: Subgroup C
Dietary Supplement: Myo-inositol plus D-chiro inositol — Myo-inositol plus D-chiro inositol 550mg/13,8 mg twice a day
  Arms: Subgroup D

SUMMARY:
The investigators aim to compare the effect of different inositol stereoisomers supplementation in lowering insulin resistance levels after 8 weeks of treatment in pregnant women with GDM and in preventing adverse obstetric outcomes.

The study population includes 80 women with GDM, randomly allocated to subgroup A (folic acid 400 mcg/day), subgroup B (myo-inositol 2000 mg twice a day), subgroup C (D-chiro-inositol 250 mg twice a day), and subgroup D (Myo-inositol plus D-chiro-inositol 550mg/13,8 mg twice a day).

Folic acid or inositol stereoisomers will be administered starting at the enrolling time (24-28 week gestation, after GDM diagnosis) till the delivery.

The homeostasis model assessment of insulin resistance (HOMA-IR) and the sensitivity index (QUICKI) will be checked at the moment of the diagnostic oral glucose tolerance test (24-28 weeks) and after 8 weeks of treatment. Obstetric outcomes, the rate of women needed insulin therapy and insulin dosage will be registered.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance that begins or is first recognized during pregnancy (1). It is characterized by an increase of physiological insulin resistance and it is associated with an increased risk of perinatal and maternal morbidity (2,3).

Inositol is a six-carbon polyol, normally present in a variety of foods, which has been classified as an insulin sensitizing agent. It exists as nine different isomers including myo-inositol (MI) and D-chiro-inositol (DCI) that are the most represented in human body. Myo-inositol and D-chiro-inositol glycans administration has been reported to exert beneficial effects at metabolic, hormonal and ovarian levels (4-5).

Recently has been demonstrated that Myo-inositol supplementation improves insulin resistance in patients with GDM (6), whereas there aren't data about the use of D-chiro-inositol or Myo-inositol plus D-chiro-inositol in women affected by GDM.

In this proposed study, the investigators aim to compare the effect of different inositol stereoisomers supplementation (Myo-inositol, D-chiro-inositol or Myo-inositol plus D-chiro-inositol ) in lowering insulin resistance levels after 8 weeks of treatment in pregnant women with GDM and in preventing adverse obstetric outcomes. All the available inositol formulations also contain folic acid (200 mcg).

The study population includes 80 women with GDM, randomly allocated to subgroup A (folic acid 400 mcg/day), subgroup B (myo-inositol 2000 mg twice a day), subgroup C (D-chiro-inositol 250 mg twice a day), and subgroup D (Myo-inositol plus D-chiro-inositol 550mg/13,8 mg twice a day).

Dietary control, folic acid or inositol stereoisomers will be administered starting at the enrolling time (24-28 week gestation, after GDM diagnosis) till the delivery.

The homeostasis model assessment of insulin resistance (HOMA-IR) and the sensitivity index (QUICKI) will be checked at the moment of the diagnostic oral glucose tolerance test (24-28 weeks) and after 8 weeks of treatment. Obstetric outcomes, the rate of women needed insulin therapy and insulin dosage will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Diabetes diagnosed within 24-28 weeks gestation
* Caucasian pregnant women

Exclusion Criteria:

* Pre-pregnancy diabetes
* Non-singleton pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance level evaluated by homeostasis model assessment of insulin resistance (HOMA-IR) | 56 days- 8 weeks

SECONDARY OUTCOMES:
hypertensive disorders | 56 days- 8 weeks
macrosomia | at delivery
cesarean section | at delivery
neonatal hypoglycemia | at delivery
jaundice requiring phototherapy | within the first 2 weeks after delivery
lipid profile | 56 days- 8 weeks
insulin therapy requirements | 56 days- 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital "SS Annunziata", Chieti, Chieti, Italy

REFERENCES:
- [Background] Metzger BE, Coustan DR. Summary and recommendations of the Fourth International Workshop-Conference on Gestational Diabetes Mellitus. The Organizing Committee. Diabetes Care. 1998 Aug;21 Suppl 2:B161-7. No abstract available. PMID 9704245
- [Background] Casey BM, Lucas MJ, Mcintire DD, Leveno KJ. Pregnancy outcomes in women with gestational diabetes compared with the general obstetric population. Obstet Gynecol. 1997 Dec;90(6):869-73. doi: 10.1016/s0029-7844(97)00542-5. PMID 9397092
- [Background] Jovanovic L, Pettitt DJ. Gestational diabetes mellitus. JAMA. 2001 Nov 28;286(20):2516-8. doi: 10.1001/jama.286.20.2516. No abstract available. PMID 11722247
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Derived] Fraticelli F, Celentano C, Zecca IA, Di Vieste G, Pintaudi B, Liberati M, Franzago M, Di Nicola M, Vitacolonna E. Effect of inositol stereoisomers at different dosages in gestational diabetes: an open-label, parallel, randomized controlled trial. Acta Diabetol. 2018 Aug;55(8):805-812. doi: 10.1007/s00592-018-1157-4. Epub 2018 May 17. PMID 29774465